CLINICAL TRIAL: NCT06114576
Title: Effects of Orange Juice Enriched With Vitamin D3 and Encapsulated Probiotics in High Cardiometabolic Risk Individuals
Brief Title: Effects of Biofunctional Orange Juice on Cardiometabolic Risk Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agricultural University of Athens (Other)
Responsible Party: Principal Investigator, Aimilia Papakonstantinou, Assistant Professor, Agricultural University of Athens
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HRPD 75/04.10.2022
Record Dates: First submitted 2023-10-18; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Overweight and Obesity; Prediabetes; Hypertension; Dyslipidemias
Keywords: orange juice; vitamin D3; probiotics; cardiometabolic risk factors
MeSH Terms: conditions — Overweight; Obesity; Prediabetic State; Hypertension; Dyslipidemias | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orange juice enriched with vitamin D3 and encapsulated probiotics (Experimental): 250 ml of orange juice enriched with vitamin D3 and encapsulated probiotics
  Interventions: Other: Orange juice enriched with vitamin D3 and encapsulated probiotics
- Conventional orange juice (Active Comparator): 250 ml of conventional orange juice
  Interventions: Other: Conventional orange juice

INTERVENTIONS:
Other: Orange juice enriched with vitamin D3 and encapsulated probiotics — 25 high cardiometabolic risk volunteers will be asked to consume 250 ml orange juice enriched with 2000 IU vitamin D3 and 10^8 cfu/ml encapsulated probiotics (Lactocaseibacillus casei shirota and Lactocaseibacillus rhamnosus GG) daily, for 8 weeks, without any other change in their dietary habits and physical activity.
  Arms: Orange juice enriched with vitamin D3 and encapsulated probiotics
Other: Conventional orange juice — 25 high cardiometabolic risk volunteers will be asked to consume 250 ml conventional orange juice daily, for 8 weeks, without any other change in their dietary habits and physical activity.
  Arms: Conventional orange juice

SUMMARY:
The effects of orange juice enriched with vitamin D3 and encapsulated probiotics (Lacticaseibacillus casei Shirota and Lacticaseibacillus rhamnosus GG) compared to conventional orange juice on several cardiometabolic and anthropometric parameters in individuals at risk of cardiovascular disease.

DETAILED DESCRIPTION:
This randomized, double-blind, controlled clinical trial aims to evaluate the effects of the consumption of orange juice enriched with vitamin D3 and encapsulated probiotics (Lacticaseibacillus casei Shirota and Lacticaseibacillus rhamnosus GG) compared to conventional orange juice in 50 high cardiometabolic risk volunteers. The participants must be overweight/obese with either prediabetes, and/or hypertension, and/or hyperlipidemia, and will be divided and randomly assigned into 2 groups of 25 individuals each. Participants will consume 250 ml of either orange juice enriched with vitamin D3 and encapsulated probiotics (Lacticaseibacillus casei Shirota and Lacticaseibacillus rhamnosus GG) or conventional orange juice daily for 8 weeks as an addition to their usual dietary intake. Participants will be asked to maintain their usual physical activity during the intervention period. At the beginning of the study and at 8 weeks, blood samples will be collected after 12 hours of fasting. Two-hour oral glucose tolerance test (OGTT) will be performed using a continuous glucose monitoring system at the beginning and at 8 weeks. Anthropometric measurements will be performed at the beginning and every week for 8 weeks. Basal metabolic rate (BMR) and central aortic blood pressure will be measured at the beginning, 4 weeks, and 8 weeks of intervention. Fecal samples will be collected and analyzed to study gut microbiome compositob at the intervention's beginning and at 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index >= 25 kg/m2
* Prediabetes [fasting blood glucose > 100 mg/dL], or/and
* Hypertension [Systolic blood pressure (SBP) > 130 mmHg or Diastolic blood pressure (DBP) > 80 mmHg], or/and
* Hyperlipidemia [total cholesterol > 200 mg/dL, and/or LDL-C > 100 mg/dL, and/or triglycerides > 150 mg/dL]

Exclusion Criteria:

* Severe chronic disease (e.g. cardiovascular diseases, diabetes mellitus, kidney or liver diseases, endocrine conditions)
* Medication that affects glycemia such as metformin, glucocorticoids, thiazide diuretics
* Gastrointestinal disorders
* Pregnancy
* Lactation
* Alcohol abuse
* Drug dependency
* Body weight lowering medications and/or history of bariatric surgery
* Depression and other psychiatric diseases
* Cancer
* Probiotic, prebiotic, and vitamin D supplemental intake

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Change in blood glucose concentrations | 8 weeks
  Clinically significant change in blood glucose concentrations (mg/dL)

SECONDARY OUTCOMES:
Change in energy intake | 8 weeks
  Clinically significant change in energy intake (kcal/day)
Change in blood lipids | 8 weeks
  Clinically significant in triglycerides (mg/dL), total cholesterol (mg/dL), low-density lipoprotein (mg/dL), and high-density lipoprotein (mg/dL)
Change in blood insulin concentrations | 8 weeks
  Clinically significant change in blood insulin concentrations (μU/L)
Change in basal metabolic rate (BMR) | 8 weeks
  Clinically significant change in basal metabolic rate (kcal/day)
Change in central aortic blood pressure | 8 weeks
  Clinically significant change in central pressure (mmHg)
Change in body weight | 8 weeks
  Clinically significant change in body weight (kg)
Change in gut microbiome | 8 weeks
  The microbial composition in fecal samples will be measured via taxonomic profiling by 16S (V3-V4 region) ribosomal RNA gene amplicon sequencing using the MiSeq Illumina platform (v3 300bp pair-end sequencing) to identify a wide diversity of microbes

CONTACTS AND LOCATIONS:
Overall Officials: Emilia Papakonstantinou, PhD, Principal Investigator — Agricultural University of Athens
Locations (1):
- Agricultural University of Athens, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No